CLINICAL TRIAL: NCT06832111
Title: The Effect of Different Kinesio Tape Applications on Balance and Ankle Joint Position Sensation: A Randomised Controlled Study
Brief Title: Kinesio Taping Effects on Balance and Ankle Proprioception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, Assistant Profesor, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UBeykent-11
Record Dates: First submitted 2025-02-06; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Ankle Injuries; Balanced
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Since you are applying different interventions (three types of Kinesio taping) to different groups, the Parallel Assignment model is the best fit.
  The study is randomized, meaning participants are assigned to groups by chance. The primary aim is to evaluate the preventive effects of Kinesio taping on balance and proprioception, so the primary purpose is "Prevention." If the person assessing the results is blinded to the group allocations, it qualifies as Single-Blinded (Outcomes Assessor).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio Taping Application 1 (Experimental): Participants in this group will receive Kinesio Taping Application 1, a specific taping technique applied to the ankle. The intervention aims to assess its effects on joint position sense and balance over four time points: before application, immediately after, 24 hours later, and 48 hours later.
  Interventions: Other: Kinesio Taping 1
- Kinesio Taping Application 2 (Experimental): Participants in this group will receive Kinesio Taping Application 2, a different taping technique applied to the ankle. The study will evaluate its impact on proprioception and postural stability over the same four time points.
  Interventions: Other: Kinesio Taping 2
- Sham Taping (Placebo Comparator) (Placebo Comparator): Participants in this group will receive a sham Kinesio taping application, which mimics the appearance of real taping but is applied without therapeutic tension or functional support. This group will serve as a placebo control to assess whether the effects observed in the experimental groups are due to the taping method or a placebo effect.
  Interventions: Other: Sham Kinesio Taping

INTERVENTIONS:
Other: Kinesio Taping 1 — A specific Kinesio taping technique applied to the ankle to evaluate its effects on joint position sense and balance.
  Arms: Kinesio Taping Application 1
Other: Kinesio Taping 2 — A different Kinesio taping technique applied to the ankle to assess its impact on proprioception and postural stability.
  Arms: Kinesio Taping Application 2
Other: Sham Kinesio Taping — A placebo taping application that mimics the real Kinesio tape placement but lacks therapeutic tension or functional support, serving as a control condition to evaluate the true effects of the experimental interventions.
  Arms: Sham Taping (Placebo Comparator)

SUMMARY:
Ankle injuries are among the most common musculoskeletal injuries, affecting both athletes and the general population. Various methods are used to prevent such injuries, but the effectiveness of different kinesio taping applications on joint position sense and balance remains unclear. This study aims to investigate the effects of different kinesio taping techniques on proprioception and postural stability in healthy young adults. By identifying changes in balance and proprioception before injuries occur, the findings may provide clinical insights into the potential role of kinesio taping in rehabilitation and injury prevention.

DETAILED DESCRIPTION:
Ankle and foot injuries are among the most frequently observed musculoskeletal injuries, particularly in athletes and physically active individuals. Various preventive methods have been developed to reduce the risk of such injuries, including exercise programs, footwear modifications, and taping techniques. Kinesio taping (KT) is widely used to enhance proprioception, joint stability, and neuromuscular function, but its effectiveness in healthy young adults remains unclear.

This study aims to evaluate the impact of different kinesio taping applications on joint position sense and balance in healthy young adults. The ankle-foot complex is rich in mechanoreceptors and plays a crucial role in movement and postural control. However, proprioceptive deficits and balance impairments contribute to the risk of injuries such as chronic ankle instability (CAI) and lateral ankle sprains. While several studies have investigated the effects of KT in injured populations, research on its impact on proprioception and balance in uninjured individuals is lacking.

By analyzing changes in balance and proprioception among healthy participants, this study will provide valuable insights into the potential role of kinesio taping in injury prevention. Understanding these effects before an injury occurs could help refine rehabilitation strategies and improve clinical decision-making regarding the use of kinesio taping for both prevention and post-injury treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be between 18-25 years old.
* General Health: Participants must be generally healthy individuals, with no previously diagnosed chronic health conditions, musculoskeletal disorders, or history of injuries.
* Ankle Health: No ankle injuries or surgical interventions in the past six months.
* Informed Consent: Participants must voluntarily agree to participate and sign the informed consent form.

Exclusion Criteria:

* History of Injuries: Any lower extremity injury (ankle or knee) within the past year.
* Neurological Disorders: Any neurological condition that may affect balance or proprioception.
* Other Health Conditions: Presence of chronic diseases such as rheumatic diseases, diabetes, or musculoskeletal disorders that could impact the study outcomes.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-24 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Joint Position Sense Accuracy | 1 months
  This outcome will assess participants' ability to accurately reproduce a predefined ankle position. A smaller error in joint position replication indicates improved proprioception.
Balance Performance (Postural Stability) | 1 months
  Participants will perform the SEBT, where they must reach as far as possible in multiple directions while maintaining balance. The total reach distance will be recorded, and improvements indicate enhanced postural stability.

SECONDARY OUTCOMES:
Changes in Balance Performance Over Time | 1 months
  The progression of balance performance will be analyzed over multiple time points to determine how long the taping effects persist.
Proprioception Retention Effect | 1 months
  Comparison between Immediately After, 24 Hours, and 48 Hours Post-Application

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin ŞAHBAZ, Principal Investigator — Istanbul Beykent University
Locations (1):
- Istanbul Beykent University Physiotherapy Lab., Istanbul, Büyükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to privacy concerns and institutional policies, individual-level data collected during this study will not be made publicly available. However, summary results and statistical analyses will be shared through scientific publications and conference presentations.